CLINICAL TRIAL: NCT00662428
Title: Evaluation of a Guideline-based Net Care Intervention to Reduce the Duration of Inpatient Depression Treatment
Brief Title: Increasing Cost-effectiveness of Inpatient Treatment of Affective Disorders
Acronym: INCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Collaborators: German Medical Association (Other)
Responsible Party: Principal Investigator, Martin Härter, Prof. Dr. Dr., University Hospital Freiburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BÄK 06-69
Record Dates: First submitted 2008-04-15; First posted 2008-04-21 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Depressive Disorder
Keywords: cost-benefit analysis; practice guideline; inpatients
MeSH Terms: conditions — Depressive Disorder | interventions — Therapeutics

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: Symptom based discharge management
- Control (Active Comparator)
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: Symptom based discharge management — Depressive symptoms of patients are weekly assessed by Beck Depression Inventory (BDI II). Patients are discharged when BDI-score is under 20 points. Patients are treated in the same hospital for two more weeks as outpatients before being referred to outpatient care (general practitioner or specialist).
  Arms: Intervention
Other: Treatment as usual — Treatment as usual is the usual stationary depression treatment which consists of a combination of several psychopharmacological and psychotherapeutical treatments. Duration of treatment is varying widely.
  Arms: Control

SUMMARY:
The cost-effectiveness of a new, guideline oriented sequential inpatient - outpatient treatment model will be investigated. Secondary outcomes are: patient satisfaction, practitioners' satisfaction and influence on work.

DETAILED DESCRIPTION:
Great diversity concerning duration of inpatient treatment of depression in psychiatric-psychotherapeutic hospitals is often used as an argument for the possible reduction of length of stay. Yet shorter duration of inpatient treatment of depressive episodes has not been examined systematically concerning clinical outcomes and health economic consequences. In this study the cost-effectiveness of a new sequential inpatient-outpatient treatment model will be examined. The research hypothesis is that the new treatment model will be more cost-effective than treatment as usual. The design provides a randomized controlled trial (RCT) in four psychiatric-psychotherapeutic clinics with a total of 240 patients. First medical practitioners and psychologist will receive a retraining concerning guideline-based care and the new treatment model will be implemented in the hospitals. New patients admitted to one of the hospitals will then be assigned randomly to one of the two study conditions und prospectively examined at five measuring times: Condition A (control group) contains treatment as usual (individual treatment programme, discharge after remission), Condition B (intervention group) contains the sequential inpatient-outpatient treatment (guideline-based treatment, discharge after partly remission: BDI <20, outpatient treatment in the hospital and guided transfer to outpatient care).

Primary outcome is the reduction of costs of treatment in relation to reduction of symptoms. Secondary outcomes will be reduction of the depressive pathology as well as the extent of satisfaction among patients and practitioners. A total of 240 patients will be examined from admission until 12 month after discharge. Both information from the patients and the practitioners will be charged with well implemented and established instruments (psychiatric basic documentation system, BADO). A specific questionnaire will be used to measure the practitioners' satisfaction and the consequences of the sequential inpatient-outpatient treatment. To answer the main question about the cost-effectiveness analyses of central health economic outcome variables (direct and indirect costs of treatment) will be performed. This study is going to give differentiated and scientific evidence of the efficiency of a new sequential inpatient-outpatient treatment for depressive disorders. The participation of psychiatric-psychotherapeutic hospitals with different functions and structures in the public health care systems (academic medical centre, psychiatric department of general hospital, psychiatric centres) enable the evaluation of the new treatment model under diverse structural and organizational conditions.

ELIGIBILITY:
Inclusion Criteria:

* Current depressive episode at time of admission
* ICD-10 diagnosis:

  * Depressive episode, F 32.xx
  * Recurrent depressive episode, F 33.xx
* Depression is primary treatment indication
* The ability to give informed consent
* Sufficient German language skills
* Being resident sufficiently close to the hospital for being able to take part in the outpatient program
* permanent residence

Exclusion Criteria:

* Dementia
* Alcohol or drug dependence (not misuse)
* Psychotic symptoms
* Schizoaffective disorders
* Bipolar disorders
* Schizophrenia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2008-05; Primary Completion 2010-09 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Cost-effectiveness: ratio of treatment response and treatment costs | one year after discharge

SECONDARY OUTCOMES:
Symptom reduction | at discharge, 6 month after discharge, and one year after discharge
patient satisfaction | at discharge

CONTACTS AND LOCATIONS:
Overall Officials: Martin Härter, Prof. Dr. Dr., Principal Investigator — Freiburg University Medical Center, Dept. of Psychiatry and Psychotherapy; Isaac Bermejo, Dr., Principal Investigator — Freiburg University Medical Center, Dept. of Psychiatry and Psychotherapy; Lars P Hölzel, Dr., Study Chair — Freiburg University Medical Center, Dept. of Psychiatry and Psychotherapy
Locations (5):
- Germany (5):
  - Krankenhaus Hofheim, Hofheim, Hesse
  - Bezirkskrankenhaus Bayreuth, Bayreuth
  - Freiburg University Medical Center, Dept. of Psychiatry and Psychotherapy, Freiburg im Breisgau
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - Klinikum am Weissenhof, Weinsberg

REFERENCES:
- [Result] Hölzel L.P., Bermejo I. & Härter M. (2011). Geordnetes Entlassmanagement - Bewertung eines neuen Behandlungsmodells zur Verkürzung der Verweildauer bei depressiven Erkrankungen. Deutsches Ärzteblatt, 108, 1050-1051.